CLINICAL TRIAL: NCT06630286
Title: A Phase 3, Randomized, Double-blind, Active-controlled Study to Evaluate a Switch to an Oral Weekly Islatravir/Lenacapavir Regimen in People With HIV-1 Who Are Virologically Suppressed on Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF)
Brief Title: Study to Compare an Oral Weekly Islatravir/Lenacapavir Regimen With Bictegravir/Emtricitabine/Tenofovir Alafenamide in Virologically Suppressed People With HIV-1
Acronym: ISLEND-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-563-5925; 2024-514046-37 (Other: European Medicines Agency)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Blinded Phase: ISL/LEN + Placebo-to-Match (PTM) B/F/TAF (Experimental): Participants will receive an initial dose of ISL/LEN (Dose A), followed by once weekly ISL/LEN (Dose B) from Day 8 onwards up to Week 96. Participants will also receive PTM B/F/TAF once daily from Day 1 up to Week 96.
  Interventions: Drug: ISL/LEN; Drug: PTM B/F/TAF
- Blinded Phase: PTM ISL/LEN + B/F/TAF (Experimental): Participants will receive an initial dose of PTM ISL/LEN (Dose A), followed by once weekly PTM ISL/LEN (Dose B) from Day 8 onwards up to Week 96. Participants will also receive B/F/TAF (50/200/25 mg) once daily up from Day 1 up to Week 96.
  Interventions: Drug: B/F/TAF; Drug: PTM ISL/LEN
- Open- Label Extension (OLE) Phase (Experimental): After the end of Blinded Phase at Week 96, if safety and efficacy of ISL/LEN are demonstrated following review of unblinded data, all participants will be given an option to enter the open-label extension phase to receive ISL/LEN in an extension phase until ISL/LEN becomes available or until the sponsor elects to discontinue the study, whichever occurs first.
  Participants receiving ISL/LEN and PTM B/F/TAF during the blinded phase will continue to take ISL/LEN weekly.
  Participants receiving B/F/TAF and PTM ISL/LEN during the blinded phase will take an initial dose of ISL/LEN (Dose A), followed by once weekly ISL/LEN (Dose B) from Day 8 onwards.
  Interventions: Drug: ISL/LEN

INTERVENTIONS:
Drug: ISL/LEN — Tablet administered orally
  Arms: Blinded Phase: ISL/LEN + Placebo-to-Match (PTM) B/F/TAF; Open- Label Extension (OLE) Phase
Drug: B/F/TAF — Tablet administered orally
  Other Names: Biktarvy®
  Arms: Blinded Phase: PTM ISL/LEN + B/F/TAF
Drug: PTM B/F/TAF — Tablet administered orally
  Arms: Blinded Phase: ISL/LEN + Placebo-to-Match (PTM) B/F/TAF
Drug: PTM ISL/LEN — Tablet administered orally
  Arms: Blinded Phase: PTM ISL/LEN + B/F/TAF

SUMMARY:
The goal of this clinical study is to learn about the safety and efficacy of switching to once weekly tablet of islatravir/lenacapavir (ISL/LEN) regimen versus continuing standard treatment of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) in people with human immunodeficiency virus (PWH) who are virologically suppressed (HIV-1 RNA levels < 50 copies/mL) on B/F/TAF for ≥ 6 months prior to screening.

The primary objective is to evaluate the efficacy of switching to oral weekly ISL/LEN tablet regimen versus continuing B/F/TAF in virologically suppressed PWH at Week 48.

ELIGIBILITY:
Key Inclusion Criteria:

* HIV-1 RNA < 50 copies/mL for ≥ 6 months before screening, as documented by:

  1. One HIV-1 RNA < 50 copies/mL immediately preceding the 24 week period prior to screening.
  2. Within 24 weeks prior to screening, if HIV-1 RNA results are available, all levels must be < 50 copies/mL.
  3. During the 6 to 12 months period prior to screening, transient detectable viremia ≥ 50 copies/mL is acceptable ("blip"), as long as it is not confirmed on 2 consecutive visits.
* Plasma HIV-1 RNA levels < 50 copies/mL at screening.
* Individuals are receiving B/F/TAF for ≥ 6 months prior to screening and willing to continue until Day 1.
* Individuals assigned female at birth and of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified methods of contraception.

Key Exclusion Criteria:

* Prior virologic failure.
* Prior use of, or exposure to ISL or LEN.
* Active, serious infections requiring parenteral therapy within 30 days before randomization.
* Active tuberculosis infection.
* Acute hepatitis within 30 days before randomization.
* Hepatitis B virus (HBV) infection as determined below at the screening visit:

  1. Positive HBV surface antigen OR
  2. Positive HBV core antibody and negative HBV surface antibody. Note: individuals found to be susceptible to HBV infection (eg negative hepatitis B surface antibody at the screening visit, regardless of prior HBV vaccination history) should be recommended to receive HBV vaccination.
* Active hepatitis C virus (HCV) coinfection, defined as detectable HCV RNA. Note: individuals with prior/inactive HCV infection (defined as undetectable HCV RNA) may be enrolled.
* Any of the following laboratory values at screening:

  1. Creatinine clearance (CLcr) ≤ 30 mL/min according to the Cockcroft-Gault formula
  2. Alanine aminotransferase > 5 x upper limit of normal (ULN)
  3. Direct bilirubin > 1.5 x ULN
  4. Platelets < 50,000/μL
  5. Hemoglobin < 8.0 g/dL

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Determined by the United States (US) Food and Drug Administration (FDA)-Defined Snapshot Algorithm | Week 48

SECONDARY OUTCOMES:
Proportion of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 96 as Determined by the US FDA-Defined Snapshot Algorithm | Week 96
Proportion of Participants with HIV-1 RNA < 50 Copies/mL at Weeks 48 as Determined by the US FDA-Defined Snapshot Algorithm | Week 48
Proportion of Participants with HIV-1 RNA < 50 Copies/mL at Weeks 96 as Determined by the US FDA-Defined Snapshot Algorithm | Week 96
Change From Baseline in Cluster of Differentiation 4 (CD4) T-Cell Count at Weeks 48 | Week 48
Change From Baseline in CD4 T-Cell Count at Weeks 96 | Week 96
Proportion of Participants Discontinuing ISL/LEN due to Treatment-Emergent Adverse Events (TEAEs) | Day 1 up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (106):
- United States (60):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pueblo Family Physicians, Phoenix, Arizona
  - Kaiser Permanente Southern California, Los Angeles, California
  - Ruane Clinical Research Group, Inc, Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - BIOS Clinical Research, Palm Springs, California
  - Optimus Medical Group, San Francisco, California
  - Vivent Health, Denver, Colorado
  - University of Colorado- Anschutz Medical Campus - PPDS, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - CAN Community Health, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - CAN Community Health, Miami Gardens, Florida
  - Midland Research Group, Inc., Oakland Park, Florida
  - Orlando Immunology Center, Orlando, Florida
  - AHF (AIDS Healthcare Foundation) - Pensacola Research, Pensacola, Florida
  - CAN Community Health, Sarasota, Florida
  - St. Josephs Comprehensive Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University, Macon, Georgia
  - Chatham CARE Center, Savannah, Georgia
  - Howard Brown Health, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - The Brigham and Women's Hospital, Inc., Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Community Research Initiative, Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Trinity Health, Grand Rapids, Michigan
  - KC CARE Health Center, Kansas City, Missouri
  - ID CARE, Hillsborough, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - AXCES Research Group - Albuquerque, Santa Fe, New Mexico
  - Brooklyn Clinical Research Center, Brooklyn, New York
  - New York Presbyterian Hospital, Flushing, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - CTRC University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Infectious Disease Kenilworth, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Brody School of Medicine at East Carolina University Adult Specialty Care, Greenville, North Carolina
  - Rosedale Health and Wellness, Huntersville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Prisma Health/USC, Columbia, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - AXCES Research Group, LLC, El Paso, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - The Crofoot Research Center, INC., Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - AXCES Research Group, LLC, Salt Lake City, Utah
  - Clinical Alliance for Research & Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
  - Peter Shalit MD, Seattle, Washington
  - MultiCare Institute for Research & Innovation, Spokane, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin
- Argentina (2):
  - Fundacion Huesped, Buenos Aires
  - Helios Salud S.A., Buenos Aires
- Australia (5):
  - East Sydney Doctors, Darlinghurst, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Surry Hills, New South Wales
  - Monash Health, Clayton, Victoria
  - Prahran Market Private Clinic, South Yarra, Victoria
- Canada (3):
  - Clinique de médecine Urbaine du Quartier Latin, Montreal
  - McGill University Health Centr, Montreal
  - Spectrum Health, Vancouver
- France (4):
  - CHU Bordeaux - Hopital Saint André, Bourdeaux
  - AP-HP-Hopital Bicétre, Le Kremlin-Bicêtre
  - Assistance Publique Hopitaux de Marseille - Hopital Sainte Marguerite, Marseile
  - CHU Nice - Hopital Archet I, Nice
- Germany (5):
  - EPIMED GmbHGesellschaft fur klinische und epidemiologische Forschung in Berlin, Berlin
  - University Hospital Bonn, Medizinische und Poliklink I, Immunologische Studienambulanz, Bonn
  - Uniklinik Kéin, Innere Medizin |, Klinisches Studienzentrum Infektiologle, Clinical Trials Unit for Infectious Diseases(CTU-ID), ISZ Geb. 80, Cologne
  - Universitatsmedizin Essen, Universitatsklinikum Essen, Klinik Dermatologie, Venerologie und Allergologie,, HPSTD-Ambulanz, Essen
  - ICH Study Center GmbH & Co.KG, Hamburg
- Japan (7):
  - Chiba University Hospital, Chiba
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - University of the Ryukyus Hospital, Okinawa
  - Osaka City General Hospital, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka Fu
  - Tokyo Medical University Hospital, Tokyo
  - Japan Institute for Health Security National Center for Global Health and Medicine, Tokyo
- Puerto Rico (2):
  - Clinical Research Puerto Rico, San Juan, PR
  - University of Puerto Rico School of Medicine, San Juan, PR
- Spain (4):
  - Complexo Hospitalario Universitario da Coruna, A Coruña
  - Hospital Universitario Vall d' Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario Regional de Malaga, Málaga
- Switzerland (3):
  - Inselspital, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Universitaetsspital Zuerich, Zurich
- Taiwan (5):
  - Kaohsuing Medical University Hospital, Kaohsiung City
  - Kaohsuing Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taoyuan General Hospital, Taoyuan
- United Kingdom (6):
  - Hawthorn House, Birmingham Heartlands Hospital (University Hospitals Birmingham NHS Foundation Trust), Birmingham
  - Clinical Research Facility (University Hospitals Sussex NHS Foundation Trust), Brighton
  - Grahame Hayton Unit, Ambrose King Centre, Royal London Hospital (Barts Health NHS Trust), London
  - Royal Free Hospital (Royal Free London NHS Foundation Trust), London
  - Clinical Research Facility, 1st Floor, St Stephen's Centre, Chelsea and Westminster Hospital (Chelsea and Westminster Hospital NHS Foundation Trust), London
  - Mortimer Market Centre (Central and North West London NHS Foundation Trust), London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06630286